CLINICAL TRIAL: NCT05372549
Title: Correlation of Oxidative Stress and Oocyte Quality in Fertility Preservation
Acronym: Ooxyd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Ovo (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IIS-1022
Record Dates: First submitted 2022-05-02; First posted 2022-05-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Fertility Preservation
MeSH Terms: interventions — Oxidative Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oncology preservation (Other)
  Interventions: Other: Oxidative stress; Other: cf-DNA; Other: MAGENTA AI
- Social (elective) preservation (Other)
  Interventions: Other: Oxidative stress; Other: cf-DNA; Other: MAGENTA AI

INTERVENTIONS:
Other: Oxidative stress — Oxidative stress occurs as soon as there is an imbalance between pro- / antioxidants, and molecules exhibiting antioxidant properties are at the forefront of fertility treatment and preservation. Oxidated stress will be measured by blood sample
Other: cf-DNA — cfDNA, extracted from blood plasma in samples collected will uncover the potential role of cfDNA as a stress signal released in response to oxidative stress
Other: MAGENTA AI — Non-invasive technique analyzing images of oocytes that can differentiate oocytes with a higher reproductive potential reflective of their quality

SUMMARY:
Whether it is for oncology or personal reasons, fertility preservation allows participants to preserve their oocytes (eggs) at their current age and condition for a better chance of having a baby in the future.

In order to proceed with fertility preservation, participants will need to undergo in vitro fertilization (IVF), which is standard practice, and take stimulation medication to stimulate production of more follicles.

The combination of both Rekovelle and Menopur for fertility preservation may increase ovarian response to stimulation and increase the number of oocytes retrieved to give better chances of embryos once the oocytes will be fertilized.

The goal in this study is to understand the effect of oxydative stress on the quality of oocytes.

For the purpose of the study and to evaluate this connection, serum levels of oxidative stress and cf-DNA in your blood will be measured.

Oocyte quality will also be assessed with Magenta, a prediction tool utilizing artificial intelligence (AI). This method is non-invasive and has no risks on the oocytes.

ELIGIBILITY:
Inclusion Criteria:

- Women 18 to 37 years of age inclusively eligible for fertility preservation for either social or oncology reason

Exclusion Criteria:

* Pregnancy and lactation
* Uncontrolled thyroid or adrenal dysfunction
* Tumours of the hypothalamus or pituitary gland
* Ovarian enlargement not due to polycystic ovarian syndrome
* Gynaecological haemorrhages of unknown aetiology
* Endometriosis stage III/IV
* Use of hormonal preparations (except for thyroid medication) during the last menstrual cycle
* Use of Coenzyme Q10 during the stimulation cycle
* Renal and/or hepatic impairment
* Hypersensitivity to any active ingredient or excipients in follitropin delta and/or HP-hMG

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing fertility preservation for oncology or social purposes
Enrollment: 179 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the correlation between the oxidative stress and the quality of oocytes | Change from baseline oxidative stress at the end of IVF controlled ovarian stimulaition
  Serum sample measure variations of oxidation-reduction potential (ORP) with MiOXSYS analyzer and by PCR

SECONDARY OUTCOMES:
Evaluation of oocyte quality by visualization | At the end of IVF stimulation
  Oocyte quality will be measured by MAGENTA AI
Assessment of good quality oocytes | IVF stimulation cycle
  Measurement of serum estradiol levels
Number of mature oocytes retrieved | IVF stimulation cycle
  Efficacy of the combination or Rekovelle and Menopur

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Olive Fertility Centre, Vancouver, British Columbia
  - Ottawa Fertility Centre, Ottawa, Ontario
  - Clinique Ovo, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No